CLINICAL TRIAL: NCT01442298
Title: A Comparison Between an Individual Low Tourniquet Pressure Versus a Standard Pressure During Total Knee Arthroplasty. A Randomized Controlled Study
Brief Title: A Comparison Between an Individual Low Tourniquet Pressure Versus a Standard Pressure During Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charlotta Olivecrona (Other)
Responsible Party: Sponsor-Investigator, Charlotta Olivecrona, RN nurse, OR nurse, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007/757-31/1-4
Record Dates: First submitted 2011-09-02; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Complications; Arthroplasty
Keywords: bloodless field; cuff pressure; limb occlusion pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional treatment (Active Comparator): the Standard method;tourniquet pressure based on systolic blood pressure, plus a safety margin.
  Interventions: Procedure: conventional measurement method
- limb occlusion pressure(LOP) (Experimental): cuff pressure is based on limb occlusion pressure measurement
  Interventions: Procedure: Limb occlusion pressure (LOP)

INTERVENTIONS:
Procedure: Limb occlusion pressure (LOP) — The tourniquet cuff pressure were decided by measurement of limb occlusion pressure (LOP) using an automated photo plethysmographic sensor connected to a ATS 3000 tourniquet apparatus (Zimmer Sweden Inc®).
  Arms: limb occlusion pressure(LOP)
Procedure: conventional measurement method — Standard method at our department, the tourniquet cuff pressure was based on the patient's systolic blood pressure and a margin that were decided by the surgeon.
  Arms: conventional treatment

SUMMARY:
The use of bloodless field is a helpful and important method in orthopedic surgery. The surgery can be done without interrupting bleedings, while keeping an exact overlook of the anatomy. However the method is not without risks, and complications of various kind may occur. One of the most important factors to minimise the risk of complications, is to keep the lowest possible cuff pressure. Previous electromyography (EMG) studies have indicated neuromuscular abnormalities after bloodless field among many patients which may lead to a prolonged rehabilitation period since they cause a postoperative weakness in the muscles. Although in these studies an unnecessary high tourniquet pressures were used and the EMG tests were made 6 weeks and 6 months after the surgery.

With today's demand for fast rehabilitation, there is a need for better knowledge if lower tourniquet pressure in bloodless field surgery may lead to less neuromuscular abnormalities.

Limb Occlusion Pressure (LOP) is the tourniquet cuff pressure required to occlude the blood flow. It accounts for a patients limb and vessel characteristics and the type and fit of the tourniquet cuff. The method has developed and is now simplified, by using an automatic (plethysmographic) sensor placed on the second toe on the involved limb, and after administration of anaesthesia, and immediately before limb preparation and draping it measures the limb occlusion pressure.

When surgery starts, the cuff is inflated again; plus a safety margin based on the LOP pressure measured. The LOP method is still rarely used it has been seen as difficult and time consuming.

The primary aim of this study is to investigate whether you can reduce the used tourniquet pressure with the new LOP measurement technique and still have a adequate bloodless field; and if this will lead to any clinical difference regarding postoperative pain. The secondary aim is to investigate the difference between the test groups concerning muscle function and wound healing and if these are remaining and of clinical importance. The third aim is to study how common neuromuscular abnormalities are after the use of bloodless field with lower cuff pressures and if there are any differences between the standard method and the LOP method.

ELIGIBILITY:
Inclusion Criteria:

* Planned for total knee arthroplasty in bloodless field
* 75 year or younger

Exclusion Criteria:

* Patients unable to read and understand Swedish
* Systolic blood pressure over 200 mmHg and a girth of the thigh over 78 cm was excluded.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Cuff pressure (mmHg) | participantswill be followed for the duration of hospital stay , an expected avarage of 4-5 days
  For patients in the control group the tourniquet cuff pressure was based on the patient's systolic blood pressure and a margin that were decided by the surgeon. In the LOP group the tourniquet cuff pressure were decided by measurement of limb occlusion pressure (LOP) by using an automated photo plethysmographic sensor connected to a ATS 3000 tourniquet apparatus
Quality of bloodless field | particpants will be followed for the duration of the hospital stay, an expected avarage of 4-5 days
  Direct after surgery the surgeon rated the quality of bloodless fiels on a visual analog scale (VAS)

SECONDARY OUTCOMES:
Postoperative pain | The participants were followed daily during their hospital stay (4-5 days) and at the two months follow up after surgery
  The patients filled in the modified WOMAC scale daily during their hospital stay. The WOMAC is a self -administered and validated health status instrument with 3 domains i.e. pain , physical function and stiffness.A wound control was performed by a ward nurse at discharged. The functional assessment included measurement of the range of motion of the knee joint and a straight leg lifting test (with 1kg weigth) and was performed at third postoperative day by an independent physiotherapist. All patients were followed up two months postoperatively (wound, ROM and WOMAC).
Range of motion (ROM) | The participants were examined at third postoperative day and at the two months follow up after surgery
Postoperative wound complications | The participants were examined at discharged (day 4 or 5 postoperatively) and at the two months follow up after surgery
EMG/EnEG | Participans were examined day three and two months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of clinical science and education, Södersjukhuset, Stockholm, Sweden